CLINICAL TRIAL: NCT03062592
Title: Effects of a Naturally Occurring Dual FFAR Agonist on Incretins, Insulin Secretion, Lipids and Inflammation in Obesity and Type 2 Diabetes
Brief Title: FFAR Agonist on Incretins, Insulin, Lipids and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karina Vejrum Sørensen, MSc, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PINO2
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Type2 Diabetes Mellitus; Obesity
Keywords: incretin; insulin; glucose; appetite; ghrelin
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Subjects complete three oral glucose tolerance test (OGTT) on different days, with a minimum of one week in between. First visit is a combined screening and baseline OGTT, with no supplementation. The second and third visit subjects are randomly assigned to either 1 g of non-hydrolyzed pine nut oil or 1 g of hydrolyzed pine nut oil.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Screening/Baseline (No Intervention): A standard OGTT with no supplementation/intervention
- Non-hydrolyzed pine nut oil (Experimental): Standard OGTT supplemented with 3 g of non-hydrolyzed pine nut oil
  Interventions: Dietary Supplement: Pine nut oil
- hydrolyzed pine nut oil (Experimental): Standard OGTT supplemented with 3 g of hydrolyzed pine nut oil
  Interventions: Dietary Supplement: Pine nut oil

INTERVENTIONS:
Dietary Supplement: Pine nut oil — Subjects are supplemented with either no oil, hydrolyzed oil or non-hydrolyzed oil in combination with an OGTT
  Arms: Non-hydrolyzed pine nut oil; hydrolyzed pine nut oil

SUMMARY:
Several free fatty acids receptors (FFARs) have been discovered. These have been implicated in metabolic processes and inflammation. Consequently, these receptors have attracted interest as targets for the treatment of metabolic and inflammatory diseases, including obesity and T2D. Two of these FFARs (FFAR1, FFAR4), which is activated by specific free fatty acids (FFAs), is expressed on enteroendocrine cells, pancreatic beta-cells and adipocytes. They have been linked to 1) increased GLP-1 secretion and hence the incretin-mediated increase in glucose-stimulated insulin secretion (GSIS) and suppression of glucagon secretion, 2) a direct positive effect on GSIS, 3) reduced inflammation and 4) improved insulin sensitivity. These functions and the abundance of fatty acids in food suggests that FFARs can be considered as nutrient sensing regulators of metabolism. Roux-en-Y gastric bypass (RYGB), frequently results in immediate beneficial effects on glucose metabolism and often complete remission of T2D. This may in part be explained by increased GLP-1 levels after surgery. It appears that the effect depends on nutrient delivery directly to the lower parts of the small intestine. It is possible that the RYGB effects are partly due to enteroendocrine stimulation of FFAR1 and perhaps FFAR4 by direct nutrient delivery, i.e. FFA release in the lower intestines. Pinolenic acid from pine nuts has been shown to be a potent dual FFAR1/FFAR4 agonist.

Based on these findings the investigators have planned a number of human intervention studies in order to investigate 1) the optimal oral formulation of pine nut oil 2) whether it is possible to mimic the beneficial effects observed after RYGB, 2) if it is possible to increase meal-related GLP-1 secretion by stimulating FFAR1/FFAR4 on enteroendocrine cells causing improved GSIS and increased satiety and 3) enhancement of GSIS by directly stimulating FFAR1 (and perhaps FFAR4) on beta-cells.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is one of the greatest health challenges worldwide. The disease is strongly associated with obesity, and develops via pre-diabetic conditions, where insulin resistance and low-grade inflammation play an important role, to T2D, where failure of the pancreatic beta-cell to compensate for insulin resistance causes hyperglycemia. According to recent estimates, 350 million people worldwide suffer from diabetes. The disease typically leads to many years of reduced quality of life due to side complications such as cardiovascular disease (CVD), blindness, kidney failure and amputations. T2D is estimated to be the 4th leading cause of death in the Western world with 5-10 years reduced life expectancy. It is generally agreed that a healthy diet and increased physical activity are effective in preventing T2D, and also may help to achieve a better control of T2D and reduce risk of CVD. There is, however, not a general agreement as to what a healthy diet constitutes.

During the last decade, several cell surface receptors that respond to free fatty acids (FFA) have been discovered. These free fatty acid receptors (FFARs) belong to the superfamily of G protein-coupled 7-transmembrane receptors (GPRs), and have all been implicated in metabolic processes, energy expenditure and inflammation. Consequently, several of the receptors have attracted interest as potential targets for the treatment of metabolic and inflammatory diseases, including obesity and T2D.

FFAR1 (GPR40), which is activated by long-chain FFA, is highly expressed in pancreatic β-cells and increases glucose-stimulated insulin secretion (GSIS) [4]. There is evidence that FFAR1 is also expressed in intestinal enteroendocrine cells, where it promotes secretion of incretin hormones such as GLP-1 and GIP. GLP-1 is highly interesting for treatment of obesity and T2D because of its ability to increase GSIS, enhance β-cell growth, increase insulin sensitivity, reduce gastric motility, increase satiety and cause a loss of weight. The published phase II clinical trial with the selective FFAR1 agonist TAK-875 demonstrated high efficacy in reducing plasma glucose without increased incidence of hypoglycemia, and has caused considerable interest in the receptor as a new target for treatment of T2D.

FFAR4 (GPR120), which is activated by unsaturated long-chain FFA, is expressed in the gastrointestinal system, adipose tissue, and β-cells, and is reported to promote GLP-1 secretion from intestinal cells, to counteract inflammation and to increase insulin sensitivity in adipose tissue. Notably, dysfunctional FFAR4 was recently connected to the development of obesity in both mice and humans. This has considerably increased the interest on the receptor as a target for obesity and metabolic diseases. This is supported by indications that unsaturated FFA revert diet-induced hypothalamic inflammation through FFAR4, and thereby reduce body weight in diet-induced obese (DIO) mice. These FFARs are thus expressed in different tissues in the body where they potentially can affect metabolic and inflammatory conditions such as T2D and obesity.

These functions combined and the abundance of fatty acids in food suggests that FFARs can be considered as nutrient sensing regulators of metabolism.

Roux-en-Y gastric bypass (RYGB) surgery, often used to treat severe obesity, frequently results in immediate beneficial effects on glucose metabolism in T2D, often with complete remission. These effects are in part independent of the weight loss, but may be explained by a significant increase in GLP-1 levels immediately after surgery. Thus, it appears that the effect depends purely on delivery of nutrients and pancreatic juices directly to the lower parts of the ileum. Normally, FFA are rapidly absorbed in the upper parts of the gastrointestinal tract. It is therefore possible that the RYGB effects are partly due to enteroendocrine stimulation of FFAR1 and perhaps FFAR4 by direct nutrient delivery, that is FFA release in the lower intestines. A hypothesis to be investigated in this PhD project is that delivery of a specific naturally occurring polyunsaturated FFA with proven high efficacy on both FFAR1 and FFAR4 directly to the lower intestines can mimic the beneficial effects observed after RYGB with less expense and fewer adverse effects.

Delivery of a higher load of unabsorbed FFA to the distal small intestine can be achieved by taking advantage of enteric coating that dissolves at pH >6.0, which is observed in the lumen of the distal jejunum, ileum and colon, and is independent of the colonic flora. This enteric coating technology is well established for delivering drugs to the ileum and colon. The potential positive effect of this principle was recently reported in a small cohort of patients with T2D. Thus, delivery of small amounts of lauric acid (a C12 fatty acid) to the distal gut using enteric-coated pellets stimulated GLP-1 secretion and lowered postprandial glucose levels in response to meals. No chronic effects where tested in this study. Although not suggested by the authors, the increased release of GLP-1 could involve direct stimulation of FFAR1 and/or FFAR4 by lauric acid in the distal gut.

As a part of the FFARMED project supported by the Danish Council for Strategic Research, a screening of 36 relevant FFA and their ability to act as FFAR1 and FFAR4 agonists in vitro have been carried out to identify the most potent naturally occurring dual FFAR1/FFAR4 agonist for clinical studies. Of these, the polyunsaturated fatty acid (PUFA), pinolenic acid showed a significantly higher efficacy than the others, and was therefore selected for further studies. To further support this choice, the effect of pinolenic acid has been tested using a small dose (100 mg/kg) given 30 min prior to an oral glucose tolerance test (OGTT) in mice. Convincingly, purified pinolenic acid significantly improved glucose tolerance by reducing AUC-glucose, and peak-glucose levels when compared to control (corn oil). The efficacy was similar to that obtained with a pharmaceutical selective FFAR1 agonist (TUG-905). Pinolenic acid is a fatty acid contained in Siberian Pine nuts, Korean Pine nuts and the seeds of other pines. The highest percentage of pinolenic acid (~20%) is found in Siberian Pine nuts and the oil produced from them. Korean Pine nut oil given as hydrolyzed FFA, but not as TG, has been reported to increase secretion of GLP-1 and decrease appetite in overweight females. This supports previous results, and indicates that only purified pinolenic acid improved glucose metabolism in mice.

Hypotheses

As described above, the expression of FFAR1 and FFAR4 on intestinal enteroendocrine cells, pancreatic beta-cells and adipose tissue has been linked to 1) increased secretion of GLP-1 and hence the incretin-mediated increase in GSIS and suppression of glucagon secretion, 2) a direct positive effect on GSIS, 3) reduced inflammation, 4) improved insulin sensitivity and 5) increased energy expenditure. Based on the above findings, the investigators are performing a number of clinical trials using pinolenic acid derived from Siberian pine nuts as a naturally occurring dual FFAR1/FFAR4 agonist.

The investigators hypothesize that ingestion of a small amount of pinolenic acid given as enteric-coated pellets dissolved in the lower intestines will 1) increase meal-related GLP-1 secretion by stimulating FFAR1/FFAR4 on enteroendocrine cells causing improved GSIS and increased satiety, 2) enhance GSIS by directly stimulating FFAR1 (and perhaps FFAR4) on beta-cells, and 3) attenuate the low-grade inflammation seen in insulin resistant conditions such as obesity and T2D by stimulating FFAR4 on adipocytes.

Aims

To test the hypotheses, the aims of this project are to investigate:

1. The effect of enteric coated pellets of pinolenic acid (hydrolyzed pine nut oil) and placebo (corn oil) on tolerability, safety and levels of glycemia in five pilot studies of healthy individuals.
2. The acute effects of pinolenic acid on meal-induced changes in I) circulating levels of glucose, insulin, GLP-1, GIP and glucagon, II) plasma lipids and inflammatory markers, III) appetite ratings, and IV) substrate metabolism in patients with T2D and lean healthy and non-diabetic obese individuals.
3. The chronic effects of pinolenic acid given 3 times daily for 8 weeks on I) the incretin effect, II) GSIS, III) body composition, IV) lipids and inflammatory markers V) substrate metabolism and VI) markers of insulin resistance and inflammation in tissue biopsies (muscle and adipose tissue) in patients with T2D and non-diabetic obese individuals.

This registration covers the second of five planned pilot studies and investigates the difference in effect between pine nut oil and hydrolyzed pine nut oil on insulin, glucose and incretin hormones when administered acutely in combination with an oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* healthy, normal weight or overweight (BMI 18, 5-30 inclusive), normal glucose tolerance, non-smoker, no gastrointestinal diseases or operations, normal EKG, normal blood values (liver, kidneys, and hematology), normal blood pressure, no first relatives with diabetes, no prescriptive medicine, informed consent.

Exclusion Criteria:

* pregnancy, breastfeeding women, food allergies of importance, dietary supplements, special diets, weight change within 3 months, difficulties with consumption of capsules.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 4 hours
  Changes in blood after a 4hour OGTT (75 g glucose)

SECONDARY OUTCOMES:
insulin | 4 hours
  Changes in blood after a 4hour OGTT (75 g glucose)
incretins | 4 hours
  Changes in blood after a 4hour OGTT (75 g glucose)
c-peptid | 4 hours
  Changes in blood after a 4hour OGTT (75 g glucose)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen KV, Korfitzen SS, Kaspersen MH, Ulven ER, Ekberg JH, Bauer-Brandl A, Ulven T, Hojlund K. Acute effects of delayed-release hydrolyzed pine nut oil on glucose tolerance, incretins, ghrelin and appetite in healthy humans. Clin Nutr. 2021 Apr;40(4):2169-2179. doi: 10.1016/j.clnu.2020.09.043. Epub 2020 Oct 2. PMID 33059911